CLINICAL TRIAL: NCT05655559
Title: Comparison of Oxygenation of the Vastus Lateralis Muscle During Cycling and Treadmill Exercises
Brief Title: Muscle Oxygenation in Treadmill and Cycle Ergometer Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Muscle_oxygenation
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Muscle Oxygenation; Treadmill
Keywords: muscle oxygenation; treadmill; cycle; moxy; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill Group (Experimental): Hemodynamic effects such as heart rate, blood pressure, oxygen saturation (SpO2), dyspnea and fatigue including muscle oxygenation, will be compared during treadmill exercises.
  Interventions: Other: Questionnare; Device: Moxy Muscle Oxygen Monitor
- Cycle Group (Experimental): Hemodynamic effects such as heart rate, blood pressure, oxygen saturation (SpO2), dyspnea and fatigue including muscle oxygenation, will be compared during cycling exercises.
  Interventions: Other: Questionnare; Device: Moxy Muscle Oxygen Monitor

INTERVENTIONS:
Other: Questionnare — Measurement of Dyspnea and Fatigue during submaximal exercise with The Modified Borg Scale (MBS).
Device: Moxy Muscle Oxygen Monitor — Measurement of muscle oxygenation with Moxy Muscle Oxygen Monitor.

SUMMARY:
The study will be conducted on healthy young adults. Hemodynamic effects such as heart rate, blood pressure, oxygen saturation (SpO2), including muscle oxygenation, will be compared in treadmill and bicycle exercises.

DETAILED DESCRIPTION:
In recent studies, sensor systems that measure the oxygen level in muscle tissue at the microvascular level have been developed. These devices working with Near Infrared Spectroscopy (NIRS, 630-850 nm) method; It provides measurements of muscle oxygenation level at rest and during exercise. It is known that significant changes in vastus lateralis oxygenation levels measured by the NIRS method are associated with various factors such as exercise intensity, exercise profile and training. The aim of this study is to measure the oxygenation level of the vastus lateralis muscle during the exercises performed on the treadmill and bicycle ergometer, and thus to reveal the effect of using different ergometers on fatigue and sportive performance.

Muscle oxygen levels will be measured and evaluated before, during and after exertion. In addition, blood pressure (BP), oxygen saturation (SpO2), dyspnea and fatigue parameters will be recorded and evaluated. If undesirable symptoms are observed during our study, the exercise will be terminated. Within the scope of the project, the acute effect will be examined with the measurements made with the Moxy device on the vastus lateralis muscle during the treadmill and bicycle ergonometer.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* No known disease
* Be between the ages of 18-25

Exclusion Criteria:

* Having cardiopulmonary disease,
* Have had lower extremity muscle or joint injuries
* Having an orthopedic/neurological disorder
* Smoking and alcohol use,
* Have suffered a lower extremity muscle or joint injury,
* Having an orthopedic/neurological disorder,
* Uncontrollable asthma,
* PaO2< 50 mmHg,
* PaCO2> 70mmHg,
* Individuals with a resting systolic blood pressure of 200 mmHg

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of Patient-Reported Dyspnea and Fatigue | Baseline
  Measurement of dyspnea during submaximal exercise with The Modified Borg Dyspnea Scale (MBS).
Measurement of Muscle Oxygenation | Baseline
  Measurement of muscle oxygenation with Moxy Monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Esra PEHLİVAN, Assoc. Prof., Study Director — Saglik Bilimleri Universitesi

IPD SHARING:
Plan to Share IPD: No